CLINICAL TRIAL: NCT01703026
Title: Contrast Enhanced EUS Using Definity in the Evaluation of Pancreatic Cancer and Pancreatic Masses
Brief Title: Contrast Enhanced EUS in the Evaluation of Pancreatic Cancer and Pancreatic Masses
Status: Completed | Type: Observational
Sponsor: Changi General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CTC0900328
Record Dates: First submitted 2012-10-05; First posted 2012-10-10 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Contrast enhanced EUS with the sonographic contrast agent DEFINITY™ has the potential to detect pancreatic cancer at an earlier stage, to improve current method of T staging and assessment of surgical resectability and also to distinguish between benign and malignant pancreatic masses. All these will translate into better clinical outcome, and also avoid unnecessary surgery in situations of unresectable cancers.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients over a 1-year period referred for EUS examination due to suspected pancreatic lesions will be enrolled.
* Age 21 years and above.
* Ability to provide informed consent

Exclusion Criteria:

Patients with clinical conditions that preclude the use of DEFINITY™ will be excluded. These conditions are:

* Right-to-left, bi-directional, or transient right-to-left cardiac shunts;
* Worsening or clinically unstable congestive heart failure;
* Acute myocardial infarction or acute coronary syndromes;
* Serious ventricular arrhythmias or high risk for arrhythmias due to prolongation of the QT interval;
* Respiratory failure;
* Severe emphysema, pulmonary emboli or other conditions that cause pulmonary hypertension due to compromised pulmonary arterial vasculature;
* Hypersensitivity to DEFINITY™ or its components.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 50 subjects will be enrolled. The study population will be drawn from patients referred for EUS evaluation on basis of suspected pancreatic cancer. These patients could be either from clinics or from the hospital wards.
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2009-08; Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Changi General Hospital, Singapore, Singapore

REFERENCES:
- [Background] Bilimoria KY, Bentrem DJ, Ko CY, Ritchey J, Stewart AK, Winchester DP, Talamonti MS. Validation of the 6th edition AJCC Pancreatic Cancer Staging System: report from the National Cancer Database. Cancer. 2007 Aug 15;110(4):738-44. doi: 10.1002/cncr.22852. PMID 17580363
- [Background] Ang TL. Endoscopic ultrasound: moving from diagnostics to therapeutics. J Dig Dis. 2008 Aug;9(3):117-28. doi: 10.1111/j.1751-2980.2008.00333.x. PMID 18956589
- [Background] Snady H, Cooperman A, Siegel J. Endoscopic ultrasonography compared with computed tomography with ERCP in patients with obstructive jaundice or small peri-pancreatic mass. Gastrointest Endosc. 1992 Jan-Feb;38(1):27-34. doi: 10.1016/s0016-5107(92)70326-5. PMID 1612375